CLINICAL TRIAL: NCT02310386
Title: The Efficacy of the BEMER Electromagnetic Field Therapy in the Treatment of Fibromyalgia.
Brief Title: BEMER in the Treatment of Pain in Fibromyalgia.
Acronym: Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Dnro 1/2014
Record Dates: First submitted 2014-11-21; First posted 2014-12-08 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Electromagnetic field therapy; Randomized controlled trial
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- activated BEMER-device (Active Comparator): Activated BEMER electromagnetic field therapy (BEMER, Innomed International, AG, Lichtenstein).
  Interventions: Device: BEMER electromagnetic field therapy
- inactivated BEMER-device (Sham Comparator): Inactivated BEMER electromagnetic field therapy (BEMER, Innomed International, AG, Lichtenstein).
  Interventions: Device: BEMER electromagnetic field therapy

INTERVENTIONS:
Device: BEMER electromagnetic field therapy — To study the effects of three months electromagnetic field therapy on pain in women with fibromyalgia.
  Other Names: BEMER, Innomed International AG, Lichtenstein

SUMMARY:
Fibromyalgia is one the most common causes of chronic pain syndromes in women. It causes considerable costs in primary health care setting as well as specialized medical care sector.Electrotherapy and exercise therapy has shown to have short-term pain relieving effects in randomized controlled trials (RCT) among fibromyalgia patients. However, there is sparse knowledge about the effects of long-term RCTs in the treatment of pain in fibromyalgia, as there are no publications about cost-effectiveness analysis of such treatments.

The aim of this study is to investigate whether the BEMER electromagnetic field therapy device has beneficial long-term effects in the treatment of pain, and whether it improves fibromyalgia patients' quality of life. In addition, this study investigates whether the BEMER device treatment is cost-effective in the treatment of fibromyalgia patients.

DETAILED DESCRIPTION:
The participants of this study are working age female patients from the Central Finland Health Care District, and who have been treating because of severe pain. After eligibility has been assessed by health-related questionnaire and clinical examination, the participants will be randomly assigned into the treatment or control group. Treatment group patients will receive the loan activated BEMER-care unit, while controls will receive inactivated sham BEMER-unit. All participants will use the device regularly on a daily bases over three months. After one month treatment break, the treatment group will become a control group and control group will become a treatment group according cross-over design principle. Switching the groups will take place by changing the BEMER devices during the break. Throughout the study, both participants and researchers are unaware whether the participants are using activated or inactivated BEMER-devices. The research will be carried out and coordinated by Central Finland Central Hospital, and the research project will take place between September 2014 and June 2018.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia
* chronic persistent moderate or severe pain for more than 12 months
* average minimum pain intensity of 5 in the scale of 0 to 10 during the last 7 days
* age between 18 and 60 years
* female gender

Exclusion Criteria:

* an inflammatory rheumatic disease
* some other chronic pain disease as fibromyalgia
* psychiatric illness
* addiction to opiates
* substance abuse
* smoking
* a person with disability
* pregnancy and breast-feeding

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain and stiffness | Change from Baseline Pain and Stiffness at 3 months
  Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Cost-effectiveness | Three Months Before and After the Start of the Intervention
  Questions about the use of drugs, visit to doctors, physiotherapy visits, and other health-care visits.
Severity of depression | Change from Baseline Severity of Depression at 3 Months
  Depression Scale (DEPS)
Quality of life | Change from Baseline Quality of Life at 3 month
  RAND-36 Questionnaire
Symptoms and functional ability | Change from Baseline Symptoms and Functional Ability at 3 months
  Fibromyalgia Impact Questionnaire (FIQ)

OTHER OUTCOMES:
Average weekly amount of symptoms (pain, stiffness, quality of sleep, vitality) | Up to 3 months
  VAS
Number of daily treatments/drugs | Up to 3 months
  Diary

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, PhD, Principal Investigator — Central Finland Health Care District, Jyväskylä, Finland, FIN-40620
Locations (1):
- Jyväskylä Central Hospital, Jyväskylä, Central Finland, Finland